CLINICAL TRIAL: NCT04917523
Title: Immunogenicity Non-inferiority Immuno-bridging Study of Inactivated SARS-CoV-2 Vaccine in Healthy Population Aged 3-17 Years Old vs Healthy Population Aged 18 Years Old and Above
Brief Title: Immuno-bridging Study of Inactivated SARS-CoV-2 Vaccine in Healthy Population Aged 3-17 vs Aged 18 Years Old and Above
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Beijing Institute of Biological Products Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CNBG2021001
Record Dates: First submitted 2021-06-04; First posted 2021-06-08 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: COVID-19 Pneumonia; COVID-19
Keywords: SARS-CoV-2; SARS-CoV-2 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Aged 3-6 years old (Experimental): 300 subjects receive 2 dose according to the immunization schedule of D0, D21 (+7 Days). A booster dose might be introduced.
  Interventions: Biological: SARS-CoV-2 Vaccine (Vero Cell), Inactivated
- Aged 7-12 years old (Experimental): 300 subjects receive 2 dose according to the immunization schedule of D0, D21 (+7 Days). A booster dose might be introduced.
  Interventions: Biological: SARS-CoV-2 Vaccine (Vero Cell), Inactivated
- Aged 13-17 years old (Experimental): 300 subjects receive 2 dose according to the immunization schedule of D0, D21 (+7 Days). A booster dose might be introduced.
  Interventions: Biological: SARS-CoV-2 Vaccine (Vero Cell), Inactivated
- Aged ≥18 years old (Active Comparator): 300 subjects receive 2 dose according to the immunization schedule of D0, D21 (+7 Days). A booster dose might be introduced.
  Interventions: Biological: SARS-CoV-2 Vaccine (Vero Cell), Inactivated

INTERVENTIONS:
Biological: SARS-CoV-2 Vaccine (Vero Cell), Inactivated — 0.5 mL per dose, containing 6.5U inactivated SARS-CoV-2 antigen

SUMMARY:
This is a open label clinical trial to evaluate the efficacy, safety and immunogenicity of inactivated SARS-CoV-2 vaccines (Vero cell) in healthy people aged 3-17 years old in comparison with healthy population aged 18 years old and above

DETAILED DESCRIPTION:
This is a open label clinical trial to evaluate the efficacy, safety and immunogenicity of inactivated SARS-CoV-2 vaccines (Vero cell) developed by Beijing Institute of Biological Products Co., Ltd in healthy people aged 3-17 years old in comparison with healthy population aged 18 years old and above. Total of 1800 healthy volunteers aged 3 years old and above will be enrolled, of whom the subjects will be divided into two groups, 3-17 years old group and 18 years old and above group with each consisting of 900 volunteers. The 3-17 years old group was further divided into three subgroups: 3-6 years old, 7-12 years old and 13-17 years old, with 300 volunteers in each subgroup. 2 doses of vaccines will be injected into the deltoid muscle of either upper arm according to the immunization schedule of D0, D21 (+7 Days). Based on interim analysis'results of the booster dose administered to adults aged 18 years old and above, a booster dose might be introduced.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 3 years old and above
* Medical history and physical examination of the subject confirms the subject is in a healthy condition and is approved by the investigator
* Female subjects of childbearing age who are not nursing or pregnant at the time of enrolment (negative urine pregnancy test) and have no family planning within the first 3 months after enrolment. Effective contraceptive measures have been taken within 2 weeks before inclusion.
* The subject must be able and willing to complete the whole immunization schedule of the study and be able to follow up study procedures for 6 months.
* With self-ability to understand the study procedures, the informed consent & voluntarily sign an informed consent/ assent form. Legal authority or parents/guardians of minors 3-17 years should sign an informed consent form and be able to comply with the requirements of the clinical study protocol.

Exclusion Criteria:

* Confirmed acute cases of SARS-CoV-2 infection.
* With a medical history of SARS, MERS virus infection (self-report, on-site inquiry);
* Fever (axillary temperature > 37.0 ℃), dry cough, fatigue, nasal obstruction, runny nose, pharyngeal pain, myalgia, diarrhea, shortness of breath and dyspnea within 14 days before vaccination (Tympanic temperature / Temporal artery temperature >37.5 ℃);
* Positive urine pregnancy test result.
* Body temperature axillary ≥ 37.0 ℃ before vaccination（Tympanic temperature / Temporal artery temperature≥ 37.5 ℃);
* With previous severe allergic reactions (such as acute allergic reactions, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain) or allergy to known ingredients of the inactivated SARS-CoV-2 vaccine.
* With a medical history or a family history of convulsion, epilepsy, encephalopathy or mental illness.
* With congenital malformation or developmental disorder, genetic defects, severe malnutrition, etc.;
* With known or suspected diseases include acute respiratory diseases (e.g. influenza like illness, acute cough, sore throat), severe cardiovascular diseases, severe liver diseases, severe kidney diseases, uncontrollable hypertension (systolic blood pressure > 150 mmHg, diastolic blood pressure > 90 mmHg), diabetic complications, malignant tumors, various acute diseases, or acute attack period of chronic diseases.
* Has been diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases; With a history of coagulation dysfunction (such as coagulation factor deficiency, coagulation disease);
* With a history of coagulation dysfunction (such as coagulation factor deficiency coagulation disease);
* Receiving anti-TB therapy.
* Receiving immune enhancement or inhibitor therapy within 3 months (continuous oral or IV administration for more than 14 days);
* Vaccinated live attenuated vaccine within 1 month before vaccination and other vaccines within 14 days before vaccination;
* Received blood products within 3 months before vaccination;
* Received other investigational drugs within 6 months before vaccination;
* Other circumstances judged by investigators that were not suitable for participating in this clinical trial.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1800 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
The four-fold increase rate of anti-SARS-CoV-2 neutralizing antibody | 28 days after 2 dose of immunization
  ≥4 fold increase from baseline
The Geometric Mean Titer (GMT) of anti-SARS-CoV-2 neutralizing antibody | 28 days after 2 dose of immunization
  Neutralizing antibody assay will be performed using the Microcytopathic assay

SECONDARY OUTCOMES:
Safety index-Incidence of adverse reactions | From the beginning of the vaccination to 28 days after the full course immunization
  the adverse event at injection site and systemic adverse event and other adverse events of the subjects are actively followed up and recorded in the subject diary card or follow-up calls
Safety index-Incidence of serious adverse events | From the beginning of the vaccination to 6 months after the full course immunization
  All SAEs will be collected
The four-fold increase rate of anti-SARS-CoV-2 neutralizing antibody | 28 days after booster dose of immunization
  ≥4 fold increase from baseline
The Geometric Mean Titer (GMT) of anti-SARS-CoV-2 neutralizing antibody | 28 days after booster dose of immunization
  Neutralizing antibody assay will be performed using the Microcytopathic assay
The distribution of neutralizing antibody titer | 28 days after 2 dose of immunization and booster dose
  The proportions of neutralizing antibody titer

CONTACTS AND LOCATIONS:
Overall Officials: Nawal Al Kaabi, MD, Principal Investigator — Sheikh Khalifa Medical City
Locations (1):
- Sheikh Khalifa Medical City, SEHA, Abu Dhabi, United Arab Emirates